CLINICAL TRIAL: NCT05325216
Title: Urinary Continence of Female Pelvic Organ-preserving Radical Cystectomy and Orthotopic Ileal Neobladder: A Randomized Controlled Study
Brief Title: Urinary Continence of Female POPRC and OIN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-KY-074
Record Dates: First submitted 2022-04-05; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Urinary Bladder Neoplasms; Woman; Sexual Dysfunction, Physiological; Treatment Outcome; Urinary Incontinence
Keywords: Bladder cancer, Female, Pelvic organ preserving-radical cystectomy, Radical cystectomy, Orthotopic ileal neobladder
MeSH Terms: conditions — Urinary Bladder Neoplasms; Sexual Dysfunction, Physiological; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POPRC group (Experimental): pelvic-organ preserving radical cystectomy with orthotopic ileal neobladder
  Interventions: Procedure: POPRC+OIN
- SRC group (Active Comparator): standard radical cystectomy with orthotopic ileal neobladder
  Interventions: Procedure: SRC+OIN

INTERVENTIONS:
Procedure: POPRC+OIN — Pelvic-organ preserving radical cystectomy with orthotopic ileal neobladder
  Arms: POPRC group
Procedure: SRC+OIN — Standard radical cystectomy with orthotopic ileal neobladder
  Arms: SRC group

SUMMARY:
To compare the urinary continence rate and long-term oncological outcomes of pelvic-organ preserving radical cystectomy (POPRC) with orthotopic ileal neobladder (OIN) versus standard radical cystectomy(SRC) with OIN.

DETAILED DESCRIPTION:
Radical cystectomy is the gold standard for muscle-invasive bladder. Orthotopic ileal neobladder, as one of the urinary diversion methods, is preferred whenever possible to achieve a better postoperative quality of life.

For standard radical cystectomy (SRC) in females, the uterus, fallopian tubes, ovaries, anterior vaginal wall, and regional lymph nodes undergo en bloc resection with the bladder and urethra . With regard to the wide range of resection, continence disorder and sexual dysfunction are very common after surgery. Pelvic-organ sparing radical cystectomy involves the preservation of the female vagina, uterus, neurovascular bundles, and any enhancement of the aforementioned techniques . Previous studies demonstrated that POPRC might not affect long-term survival and instead improve continence outcomes. However, most of the available studies are retrospective with limited cases in a single center. The current study primarily aims to urinary continence rate and long-term oncological outcomes of POPRC+OIN versus SRC+OIN in a prospective randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged between 55-75.
2. Patients those who are diagnosed with organ-confined urothelial carcinoma（<pT3）
3. Patients those who are capable for radical cystectomy with orthotopic ileal neobladder.
4. ECOG score between 0-2;
5. Normal renal function;
6. Patients those who volunteer to participate in this study and sign the informed consents.
7. Patients those who are able to cooperate in the study.

Exclusion Criteria:

1. Absence of tumour in bladder neck or urethra;
2. Patients thsoe who are diagnosed distant metastasis before surgery.
3. Previous history of malignancy of pelvic organs or surgical resection of pelvic organs;
4. Patients those who are diagnosed with other malignancies.;
5. Patients those who had received pelvic radiotherapy or major pelvic operation.
6. Pregnancy status;
7. Any other conditions that the researcher considers to be excluded from this study

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
day-time and night-time continence rate | 6 months
  We will use pad-test to evaluate the urinary continence for patients

SECONDARY OUTCOMES:
postoperative sexual function | 6 months
  International index of erectile function-5 (IIEF-5)
perioperative complications rate | 1 months
  perioperative complications rate within 1 month
overall survival | 5 years
  5-year overall survival rate
recurrence-free survival | 5 years
  5-year overall recurrence-free survival rate
operative time | 24 hours
  operative time (mins)
estimated blood loss | 24 hours
  estimated blood loss (ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
IPD will be public access via the ResMan